CLINICAL TRIAL: NCT04227002
Title: Clinical Cohort Study - Hamburg AoRtic Valve cOhoRt
Brief Title: Hamburg AoRtic Valve cOhoRt
Acronym: HARbOR
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: HARbOR
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

SUMMARY:
The primary aim of the study is to identify the optimal treatment modality for patients with aortic valve disease, incorporating the individual patient's risk profile and anticipated clinical outcomes. This includes the association of demographic factors, procedural data and biomarkers with clinical outcome in a prospective fashion.

DETAILED DESCRIPTION:
Patients with severe aortic valve disease have a poor prognosis under medical therapy, making replacement of the failing valve the preferred option. In addition to surgical aortic valve replacement (SAVR), transcatheter aortic valve implantation (TAVI) has evolved as an alternative treatment option for patients at intermediate and high operative risk. Before expansion of TAVI to low-risk and younger patients can be recommended, several questions remain to be investigated, e.g. optimal patient selection, periprocedural complications and long-term durability. Therefore every patient with a relevant aortic valve disease (aortic stenosis, aortic regurgitation or degenerative aortic valve prosthesis) who meets the inclusion/exclusion criterias is planned to be involved in the study.

Predictors of outcome are yet to be defined in patients with aortic valve disease in order to improve risk prediction for the different treatment modalities (medical, SAVR, TAVI).

The primary aim of the study is to identify the optimal treatment modality for the individual patient, incorporating the individual patient's risk profile and anticipated clinical outcomes. This includes the association of demographic factors, procedural data and biomarkers with clinical outcome in a prospective fashion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically relevant aortic valve disease (aortic valve stenosis, aortic regurgitation, degenerated aortic valve prosthesis)
* Written informed consent

Exclusion Criteria:

* Insufficient knowledge of the German language (able to understand and write the German language)
* Physical or psychological incapability to take part in the investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The medical condition being studied is aortic valve disease
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2039-09-01 (Estimated); Study Completion 2049-09-01 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | one year
  The primary aim of the study is to investigate all cause mortality after surgical aortic valve replacement or transcatheter aortic valve replacement. Events of death will be registered either from in-house information or telephone follow-up of the patient or the referring physician as part of clinical routine.

SECONDARY OUTCOMES:
Myocardial Infarction | 30 days after index procedure
  Myocardial infarction based on a combination of clinical criteria, ecg changes indicative of new ischemia and a significant rise in cardiac biomarkers (peak value exceeding 15 x as the upper reference limit for troponin or 5 x for CK-MB) within the first 72 hours (periprocedural myocardial infarction) or 30 days (spontaneous myocardial infarction) after index procedure
Stroke | 30 days after procedure
  Assessment of clinical disability using a modified Rankin Scale (mRS) within the first 30 days after index procedure
Vascular complications and bleeding | 30 days after procedure
  Evaluation of overt bleeding or vascular complications after index procedure by drop in haemoglobin and transfusion of packed red blood cells
Durability of the implanted aortic valve prosthesis | 10 years
  Evaluation of long time durability of the implanted aortic valve prosthesis by echocardiography in the yearly follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Moritz Seiffert, MD, Principal Investigator — University Heart Center Hamburg
Locations (1):
- Universitäres Herz- und Gefäßzentrum, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Westermann D, Ludwig S, Kalbacher D, Spink C, Linder M, Bhadra OD, Nikorowitsch J, Waldschmidt L, Demal T, Voigtlander L, Schaefer A, Seiffert M, Pecha S, Schofer N, Greenbaum AB, Reichenspurner H, Blankenberg S, Conradi L, Schirmer J. Prevention of coronary obstruction in patients at risk undergoing transcatheter aortic valve implantation: the Hamburg BASILICA experience. Clin Res Cardiol. 2021 Dec;110(12):1900-1911. doi: 10.1007/s00392-021-01881-4. Epub 2021 Jun 22. PMID 34156524